CLINICAL TRIAL: NCT02846103
Title: Study of Anti-telomerase T CD4 Immunity in Metastatic Lung Cancer
Acronym: Telocap02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P/2013/207
Record Dates: First submitted 2016-07-13; First posted 2016-07-27 (Estimated); Last update posted 2023-09-18 (Actual); Status verified 2022-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biological samples (Experimental): Blood samples will be collected at baseline, after the first-line therapy and at 12 months.
  Tumor tissues will be collected if available.
  Interventions: Other: Biological samples

INTERVENTIONS:
Other: Biological samples — blood and tumor tissue samples

SUMMARY:
Increasing evidence suggests that immune responses might be a determining factor in lung cancer tumor progression.

The impressive clinical responses obtained with immune checkpoint inhibitors (anti-PD-1/PDL-1, anti-CTLA-4) indicate that the presence of preexisting antitumor immune response is required for their efficacy and highlight the critical role of antitumor T cell immunity. Recent progress on the fields of tumor immunology underlines the critical role of CD4 helper 1 T lymphocyte (TH1) in the control of innate and adaptive anticancer immunity. Therefore, monitoring tumor specific TH1 response could be relevant in cancer patients.

In order to monitor tumor-specific CD4 Th1 responses in most cancer patients, the investigators group have previously described novel promiscuous peptides (referred as UCP:Universal Cancer Peptides) derived from human telomerase (TERT), a prototype of shared tumor antigen.

By using UCP-based immuno-assay, pre-existing UCP-specific Th1 responses have been detected in the blood of lung cancer patients (Telocap01). The frequency and magnitude of this response were inversely correlate to the disease stage. Furthermore, UCP-specific responses were significantly found in patients with low PD1+ and TIM3+ T cells.

Then in TeloCap02 study, UCP specific Th1 immune responses will be evaluated in lung cancer before and after treatment (chemotherapy, immunotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC (Non Small Cell Lung Cancer) or SCLC (small cell lung cancer)
* stade IIIb or metastatic
* Patient candidate to a first-line therapy
* Performance status 0, 1 or 2 on the ECOG scale
* Written informed consent

Exclusion Criteria:

* History of adjuvant chemotherapy for lung cancer treatment
* Patients under chronic treatment with systemic corticoids or other immunosuppressive drugs (prednisone or prednisolone ≤ 10 mg/day is allowed)
* Prior history of other malignancy except for: basal cell carcinoma of the skin, cervical intra-epithelial neoplasia and other cancer curatively treated with no evidence of disease for at least 5 years
* Active autoimmune diseases, HIV, hepatitis C or B virus
* Patients with any medical or psychiatric condition or disease,
* Patients under guardianship, curatorship or under the protection of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
overall survival | date of death from any cause (within 2 years after the initiation of the treatment)
  time between the date of initiation of treatment and the date of death from any cause

SECONDARY OUTCOMES:
UCP-specific Th1 responses measured by ELISPOT assay | up to 12 months
Progression free survival | date of first progression of the disease (within 2 years after the initiation of the treatment)
  time interval between the date of initiation of treatment and the date of first progression (local, remote [extent of the disease by RECIST v1.1] second cancer) or death from any cause.
quality of life related to health measured by EORTC-QLQC30 and LC13 questionaries. | from the inclusion to patient death, up to 2 years

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Centre Hospitalier Régional Universitaire de Besançon, Besançon
  - CHU de Dijon, Dijon
  - Centre Georges François Leclerc, Dijon
  - Institut Jean Godinot, Reims
  - Hôpitaux Universitaires de Strasbourg, Strasbourg

REFERENCES:
- [Background] Godet Y, Fabre E, Dosset M, Lamuraglia M, Levionnois E, Ravel P, Benhamouda N, Cazes A, Le Pimpec-Barthes F, Gaugler B, Langlade-Demoyen P, Pivot X, Saas P, Maillere B, Tartour E, Borg C, Adotevi O. Analysis of spontaneous tumor-specific CD4 T-cell immunity in lung cancer using promiscuous HLA-DR telomerase-derived epitopes: potential synergistic effect with chemotherapy response. Clin Cancer Res. 2012 May 15;18(10):2943-53. doi: 10.1158/1078-0432.CCR-11-3185. Epub 2012 Mar 8. PMID 22407833
- [Background] Godet Y, Dosset M, Borg C, Adotevi O. Is preexisting antitumor CD4 T cell response indispensable for the chemotherapy induced immune regression of cancer? Oncoimmunology. 2012 Dec 1;1(9):1617-1619. doi: 10.4161/onci.21513. PMID 23264913